CLINICAL TRIAL: NCT04429334
Title: Efficacy and Safety Study Exploring Nangibotide Treatment in COVID-19 pAtients With ventiLatory Support (ESSENTIAL) A Randomized, Double-blind, Placebo-controlled Study With Adaptive Features
Brief Title: Efficacy and Safety Study of Nangibotide in Patients With COVID-19 Receiving Ventilatory Support
Acronym: ESSENTIAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Inotrem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOT-C-204
Record Dates: First submitted 2020-05-29; First posted 2020-06-12 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19 | interventions — nangibotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- nangibotide (Experimental): Continuous infusion of experimental agent for up to 120 hours
  Interventions: Drug: nangibotide
- placebo (Placebo Comparator): Continuous infusion of matched placebo for up to 120 hours
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: nangibotide — nangibotide 1.0 mg/kg/h
  Arms: nangibotide
Drug: placebo — matching placebo
  Arms: placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, in which one dose of nangibotide will be tested versus placebo.

All patients with a diagnosis of COVID-19, and a requirement for respiratory support will be considered for study participation. The applicable local requirements for informed consent will be followed. Where permissible, an emergency consent procedure will be followed for patients unable to provide consent by themselves. All potential study patients will receive standard of care treatment throughout the study. Patients will receive a continuous intravenous (i.v.) infusion of nangibotide at 1.0 mg/kg/h or a matching placebo. Treatment with study drug must be initiated as early as possible but no later than 48 hours after the initiation of ventilatory support (Patients will be treated for 5 days or until discharge from critical care, whichever is sooner). Follow-up visits will be performed on days 8 and 14. The end of study visit is at day 28. A further follow up visit will be undertaken on day 60.

DETAILED DESCRIPTION:
ESSENTIAL was a randomized, double-blind, placebo-controlled trial, in which one dose of nangibotide was tested versus placebo. It took place in 14 sites in France and Belgium. The study was overseen by an independent Data Monitoring Committee (DMC).

The study was divided into two parts running sequentially without unblinding. Part 1 evaluated safety and tolerability study and included 60 patients, randomized in a 2:1 ratio of nangibotide to placebo. Part 2 included all recruited patients with an initially planned sample size of 370 patients, randomized in a 1:1 ratio of nangibotide to placebo.

All patients or their legally authorised representatives provided written informed consent or, in relevant countries, an independent physician, confirmed patient eligibility for enrolment in the trial.

Patients received a continuous intravenous infusion of nangibotide at 1.0 mg/kg/h or a matching placebo for 5 days (or until discharge from ICU, whichever was sooner). The treatment was in addition to standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Provided informed consent (emergency consent according to local regulations where approved)
2. Age 18 to 75 years (inclusive)
3. Admitted to an intensive care unit
4. Treatment with High Flow Nasal Oxygen, non-invasive ventilation or invasive mechanical ventilation for acute respiratory failure caused by COVID-19 for less than 48 hours
5. A PaO2:FiO2 ratio of <200mmHg (<26.7kPa) with a FiO2 ≥0.6
6. Confirmed laboratory diagnosis of COVID-19 within 7 days of meeting screening criteria

Exclusion Criteria:

1. Known pregnancy (positive urine or serum pregnancy test)
2. Ongoing treatment with an immunomodulatory agent not included in the standard of care for COVID-19 (including participation in clinical trials of such agents)".
3. Body mass index (BMI) ≥ 40 kg/m2or weight ≥ 130 kg
4. Anticipated transfer to another hospital, which is not a study site within 72 hours
5. Expected to die within 6 months of treatment due to underlying chronic disease
6. Limitations of care in place during current hospital admission

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events until day 28 | 28 days
  Part 1
Clinical Status (7-point Ordinal Scale) assessed at Day 28 | 28 days
  Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Garaud, MD, Study Chair — INOTREM SA
Locations (17):
- Belgium (2):
  - Clinique universitaire Saint-Luc, Brussels
  - Ziekenhuis Oost-Limburg, Genk
- France (15):
  - CHU Angers, Angers
  - Centre hospitalier Victor Dupouy, Argenteuil
  - Centre Hospitalier Germont et Gauthier, Béthune
  - CHU Dijon - Bourgogne - Hôpital François Mitterrand, Dijon
  - CHD Site la Roche sur Yon, les Oudairies, La Roche-sur-Yon
  - Centre hospitalier le Manas, Le Mans
  - Centre Hospitalier Universitaire Dupuytren, Limoges
  - Centre hospitalier de Melun, Melun
  - Hôpital Saint Eloi CHU Montpellier, Montpellier
  - Réanimation Médicale, Hôpital Central, Nancy
  - Hôpital Dieu - CHU Nanates, Nantes
  - Hôpital Cochin, Paris
  - Hôpital Civil - Nouvel Hôpital civil, Strasbourg
  - CHRU - Hôpital Bretonneau, Tours
  - Hôpital Franch-Comté Site Trevenans, Trévenans

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Francois B, Lambden S, Garaud JJ, Derive M, Grouin JM, Asfar P, Darreau C, Mira JP, Quenot JP, Lemarie J, Mercier E, Lacherade JC, Vinsonneau C, Fivez T, Helms J, Badie J, Levy M, Cuvier V, Salcedo-Magguilli M, Laszlo-Pouvreau AL, Laterre PF, Gibot S; ESSENTIAL investigators. Evaluation of the efficacy and safety of TREM-1 inhibition with nangibotide in patients with COVID-19 receiving respiratory support: the ESSENTIAL randomised, double-blind trial. EClinicalMedicine. 2023 Jun;60:102013. doi: 10.1016/j.eclinm.2023.102013. Epub 2023 May 31. PMID 37350989